CLINICAL TRIAL: NCT00987558
Title: Effect of Repeated Administration of Eslicarbazepine Acetate on the Pharmacokinetics of Simvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-124
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
Keywords: Eslicarbazepine acetate; simvastatin
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence A (Experimental): Simvastatin 80mg treatment period followed by Simvastatin 80 mg + eslicarbazepine acetate 800 mg treatment period
  Interventions: Drug: Eslicarbazepine acetate; Drug: Simvastatin
- Treatment Sequence B (Experimental): Simvastatin 80mg + eslicarbazepine acetate 800 mg treatment period followed by Simvastatin 80 mg treatment period
  Interventions: Drug: Eslicarbazepine acetate; Drug: Simvastatin

INTERVENTIONS:
Drug: Eslicarbazepine acetate
  Other Names: Zebinix
Drug: Simvastatin
  Other Names: Zocor

SUMMARY:
The primary objective was to investigate whether multiple-dose administration of ESL 800 mg once daily affects the pharmacokinetics of simvastatin, a substrate of CYP34A.

DETAILED DESCRIPTION:
This was a single centre, two-way crossover, randomised, open-label study in 24 healthy volunteers. The volunteers will receive an oral single-dose of simvastatin 80 mg on two occasions - once administered alone and once after treatment with an oral once-daily dose of 800 mg of ESL for 14 days -, separated by a washout period of 3 weeks or more

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 45 years, inclusive
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive
* Healthy as determined by pre-study medical history, physical examination, vital signs, and 12-lead ECG; negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening; clinical laboratory test results clinically acceptable at screening and admission to each treatment period;
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period
* Non-smokers or ex-smokers
* Able and willing to give written informed consent;
* If female, not of childbearing potential by reason of surgery or, if of childbearing potential, she uses one of the following methods of contraception: double barrier method: 1 male barrier method [male condom] plus 1 female barrier method (diaphragm, spermicide, or intrauterine device);
* If female, has a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders
* Clinically relevant surgical history;
* History of relevant atopy or any drug hypersensitivity (including known hypersensitivity to ESL or other carboxamide derivatives, simvastatin or other statins or any of its excipients
* History of fibromyalgia, myopathy, rhabdomyolysis or unexplained muscle pain
* Second or third-degree atrioventricular blockade not corrected with a pacemaker or any other clinically significant abnormality in the 12-lead electrocardiogram (ECG) as determined by the investigator
* History of alcoholism or drug abuse
* Consume more than 14 units of alcohol a week
* Significant infection or known inflammatory process on screening or admission to each treatment period
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period
* Use of medicines within two weeks of admission to first period that may affect the safety or other study assessments, in the investigator's opinion
* Have donated or received any blood or blood products within the 3 months prior to screening
* Vegetarians, vegans or have other medical dietary restrictions
* Cannot communicate reliably with the investigator
* Unlikely to co-operate with the requirements of the study
* Unwilling or unable to give written informed consent
* If female, is pregnant or breast-feeding
* If female, is of childbearing potential and does not use an approved effective contraceptive method (double-barrier method: 1 male barrier method [male condom] plus 1 female barrier method (diaphragm, spermicide, or intra-uterine device) or uses hormonal contraceptives
* Have received an investigational drug within 3 months of screening or is currently participating in another study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Claude Homery, MD, Principal Investigator — Biotrial, 7-9, rue Jean-Louis Bertrand, F-35000 Rennes, France
Locations (1):
- Biotrial, 7-9 rue Jean-Louis Bertrand, Rennes, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin, Then ESL + Simvastatin: Simvastatin 80 mg - Oral single-dose administered alone Washout period - 3 weeks Eslicarbazepine acetate (ESL) 800 mg - Oral once-daily dose for 14 days + Simvastatin single dose 80 mg on 14th day
- ESL, Then Simvastatin: Eslicarbazepine acetate (ESL) 800 mg - Oral once-daily dose for 14 days + Simvastatin single dose 80 mg on 14th day Washout period - 3 weeks Simvastatin 80 mg - Oral single-dose administered alone
Period: Overall Study
Arm/Group | Simvastatin, Then ESL + Simvastatin | ESL, Then Simvastatin
Started | 13 | 17
Simvastatin | 13 | 12
Washout | 13 | 12
Eslicarbazepine Acetate + Simvastatin | 13 | 17
Completed | 12 | 12
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Eslicarbazepine Acetate + Simvastatin: Simvastatin 80 mg + eslicarbazepine acetate 800 mg
  Simvastatin + ESL: Oral single-dose of simvastatin 80 mg on two occasions - once administered alone and once after treatment with an oral once-daily dose of 800 mg of ESL for 14 days - separated by a washout period of 3 weeks or more.
Arm/Group | Eslicarbazepine Acetate + Simvastatin
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Simvastatin Cmax (Maximum Plasma Concentration)
Description: Simvastatin (Reference) ESL + Simvastatin (Test)
Time Frame: Day 1 and Day 14
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Simvastatin (Reference): Simvastatin 80 mg
- ESL + Simvastatin (Test): Eslicarbazepine acetate (ESL) 800 mg + Simvastatin 80 mg
Arm/Group | Simvastatin (Reference) | ESL + Simvastatin (Test)
Number analyzed (Participants) | 24 | 24
ng/mL | 17.7 (14.0) | 6.89 (5.21)

2. Primary Outcome: Simvastatin Tmax (Time of Occurrence of Cmax)
Description: Simvastatin (Reference) ESL + Simvastatin (Test)
Time Frame: Day 1 and Day 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Simvastatin (Reference) | ESL + Simvastatin (Test)
Number analyzed (Participants) | 24 | 24
hours | 1.50 (3.29) | 1.62 (3.40)

3. Primary Outcome: Simvastatin AUC0-t
Description: AUC0-t - area under the plasma concentration versus time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification
  Simvastatin (Reference) ESL + Simvastatin (Test)
Time Frame: Day 1 and Day 14
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Simvastatin (Reference) | ESL + Simvastatin (Test)
Number analyzed (Participants) | 24 | 24
ng.h/mL | 93.9 (47.7) | 43.3 (22.5)

4. Primary Outcome: Simvastatin AUC0-∞ (AUC From Time Zero to Infinity)
Description: Simvastatin (Reference) ESL + Simvastatin (Test)
Time Frame: Day 1 and Day 14
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Simvastatin (Reference) | ESL + Simvastatin (Test)
Number analyzed (Participants) | 24 | 24
ng.h/mL | 108 (68.6) | 54.6 (46.6)

ADVERSE EVENTS:
Groups:
- Simvastatin: Simvastatin 80 mg
- Eslicarbazepine Acetate: eslicarbazepine acetate 800 mg
- Eslicarbazepine Acetate + Simvastatin: Simvastatin 80 mg + eslicarbazepine acetate 800 mg
Arm/Group | Simvastatin | Eslicarbazepine Acetate | Eslicarbazepine Acetate + Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 23/30 | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin (N=30) | Eslicarbazepine Acetate (N=30) | Eslicarbazepine Acetate + Simvastatin (N=30)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 12 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 6 | 2
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other